CLINICAL TRIAL: NCT00191685
Title: Duloxetine in the Treatment of Melancholic Depression: An 8-Week Open-Label Dose Study
Brief Title: Duloxetine in the Treatment of Melancholic Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8163; F1J-AY-HMCZ
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2006-07-25 (Estimated); Status verified 2006-07

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Duloxetine Hydrochloride

INTERVENTIONS:
Drug: duloxetine

SUMMARY:
The purpose of this study is to determine the optimal treatment strategy for MDD patients with melancholic features who do not respond to a standard daily dose. This study will allow investigators to mimic standard clinical practice. During the first 2 weeks of treatment, clinical evaluation of individual patient tolerability and efficacy will enable the dose of duloxetine to be adjusted. Patients allocated to the Flex group may have their daily dose of duloxetine adjusted in the attempt to elicit a clinical response.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of major depression with melancholic features, as defined by Diagnostic and Statistical Manual of Mental Disorders Fourth Edition [DSM-IV] criteria.
* Experienced their first episode of major depression prior to age 50.
* Have a HAMD17 total score of less than or equal to 20 at Visits 1 and 2.
* Test negative for a urine pregnancy test at Visit 1 (females).
* Agree to use medically acceptable and reliable means of birth control during the study, as determined by the investigator (females of child-bearing potential, not surgically sterilized and between menarche, and one year post-menopausal).

Exclusion Criteria:

* Have any current and primary Axis I mood disorder other than MDD, including, but not limited to, dysthymia, seasonal affective disorder or psychotic depression.
* Have a current episode of major depression that has failed to respond to two or more courses of antidepressant therapy or, in the judgment of the investigator, meets criteria for treatment-resistant depression
* Are at serious suicidal risk as determined by the investigator.
* Have a serious medical illness or clinically significant laboratory abnormalities that, in the judgment of the investigator, are likely to require medication/ intervention/ hospitalization during the course of the study.
* Had treatment with a monoamine oxidase inhibitor (MAOI) within 14 days prior to Visit 2 or potential need to use a MAOI during the study or within 14 days of discontinuation of study drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2004-05; Study Completion 2005-09

PRIMARY OUTCOMES:
To generate data to compare the proportion of outpatients with major depressive disorder with melancholic features who responded to duloxetine at a given daily dose after initially not responding to duloxetine 60mg once daily for 4 weeks.

SECONDARY OUTCOMES:
To compare outpatients with major depressive disorder with melancholic features who achieved remission after treatment with duloxetine;Collect data on the safety of duloxetine.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (23):
- Australia (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time(UTC/GMT - 5 hours, EST), or speak with your personal physician., Paddington, New South Wales
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time(UTC/GMT - 5 hours, EST), or speak with your personal physician., Everton Park, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time(UTC/GMT - 5 hours, EST), or speak with your personal physician., Hoppers Crossing, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time(UTC/GMT - 5 hours, EST), or speak with your personal physician., Nambour, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time(UTC/GMT - 5 hours, EST), or speak with your personal physician., New Farm, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time(UTC/GMT - 5 hours, EST), or speak with your personal physician., South Port BC, Queensland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time(UTC/GMT - 5 hours, EST), or speak with your personal physician., Elizabeth Vale, South Australia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time(UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Victoria
- Canada (15):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time(UTC/GMT - 5 hours, EST), or speak with your personal physician., Calgary, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time(UTC/GMT - 5 hours, EST), or speak with your personal physician., Edmonton, Alberta
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time(UTC/GMT - 5 hours, EST), or speak with your personal physician., Vancouver, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time(UTC/GMT - 5 hours, EST), or speak with your personal physician., Winnipeg, Manitoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time(UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint John, New Brunswick
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time(UTC/GMT - 5 hours, EST), or speak with your personal physician., Halifax, Nova Scotia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time(UTC/GMT - 5 hours, EST), or speak with your personal physician., Sydney, Nova Scotia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time(UTC/GMT - 5 hours, EST), or speak with your personal physician., Greater Sudbury, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time(UTC/GMT - 5 hours, EST), or speak with your personal physician., Kingston, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time(UTC/GMT - 5 hours, EST), or speak with your personal physician., London, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time(UTC/GMT - 5 hours, EST), or speak with your personal physician., Mississauga, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time(UTC/GMT - 5 hours, EST), or speak with your personal physician., Toronto, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time(UTC/GMT - 5 hours, EST), or speak with your personal physician., Beauport, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time(UTC/GMT - 5 hours, EST), or speak with your personal physician., Montreal, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 am - 5 pm Eastern Time(UTC/GMT - 5 hours, EST), or speak with your personal physician., Québec, Quebec